CLINICAL TRIAL: NCT02198885
Title: Post-marketing, Single-center, Controlled, Open-Label, Feasibility Study Comparing Use of a Prehospital Ultrasound System and Standard Prehospital Care in Patients With Thoracoabdominal Trauma.
Brief Title: Comparing Use of a Prehospital Ultrasound System and Standard Prehospital Care in Thoracoabdominal Trauma
Acronym: FAST-01
Status: Completed | Type: Observational
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatoon Health Region (Other); M.D. Ambulance Care Ltd. (Unknown)
Responsible Party: Principal Investigator, Ivar Mendez, M.D., University of Saskatchewan
Other Study IDs: FAST-01; Bio# 14-109 (Other: University of Saskatchewan Biomedical Research Ethics Board)
Record Dates: First submitted 2014-07-18; First posted 2014-07-24 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Thoracoabdominal Trauma; Focused Assessment With Sonography for Trauma (FAST); NanoMaxx Ultrasound System (SonoSite); RP-Xpress (InTouch Technologies)
Keywords: FAST; Thoracoabdominal Trauma; Prehospital care; ultrasound; NanoMaxx Ultrasound; RP-Xpress

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: This group receives the standard prehospital care en route to hospital, and they do not receive the FAST ultrasound en route.
- FAST: This group receives the FAST ultrasound en route to hospital.

SUMMARY:
The NanoMaxx Ultrasound System (SonoSite) in connection with the RP-Xpress (InTouch Technologies) provides a means of transmitting ultrasound images, video, and audio to a remote location in real-time. It has been envisioned that this system be used to diagnose trauma patients with suspected pleural effusion, hemothorax, pneumothorax, or abdominal blockage during prehospital care; under the guidance of in-hospital physicians, paramedics would perform an Focused Assessment with Sonography for Trauma (FAST) examination while trauma patients are transported to hospital via ambulance. The investigators hypothesize that in-hospital physicians interpreting ultrasound images obtained by paramedics during trauma patients' transportation to hospital will reduce time to diagnosis; thus, preparations by emergency physicians, surgeons, and operating room teams to receive critically injured patients may begin earlier, reducing time to intervention during a critical period in patient care. Data will also be collected regarding quality of images obtained in-ambulance and the interaction between paramedics and physicians using the remote-presence system.

ELIGIBILITY:
Inclusion Criteria for FAST cohort:

* Patient is 18 years of age or older
* Patient presenting with blunt or penetrating trauma to the thorax or abdomen
* Patient transported by MD Ambulance to Royal University Hospital
* Patient being transported by a paramedic who has received training in the above ultrasound system and who has with them a NanoMaxx Ultrasound System (SonoSite) to be used in connection with the RP-Xpress (InTouch Technologies)
* Patient will take longer than 10 minutes to transport to hospital
* Patient's care will not be compromised in completing a FAST exam - opinion of paramedic
* Patient's care will not be compromised in completing a FAST exam - opinion of ER physician

Inclusion Criteria for Controls:

* Patient is 18 years of age or older
* Patient presenting with blunt or penetrating trauma to the thorax or abdomen
* Patient transported by MD Ambulance to Royal University Hospital
* Patient will take longer than 10 minutes to transport to hospital

Exclusion Criteria:

* Patients under the age of 18
* Patients whose care would be compromised if other procedures of higher priority (as determined by paramedics and/or remotely-present physicians) were not be able to be executed due to time involved in completing a FAST exam
* Patients who are not being transported to Royal University Hospital
* Patients whose expected transport time from scene to hospital is less than 10 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, presenting with blunt or penetrating trauma to the thorax or abdomen, that are being transported by MD Ambulance to Royal University Hospital where the hospital trip is expected to take longer than 10 minutes.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-08; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Time to diagnosis | Within 24 hours

SECONDARY OUTCOMES:
Time to intervention | Within 24 hours

OTHER OUTCOMES:
Audio quality scores on the visual analog scale | Same day
Video quality scores on the visual analog scale | Same day

CONTACTS AND LOCATIONS:
Overall Officials: Ivar Mendez, Principal Investigator — University of Saskatchewan
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada